CLINICAL TRIAL: NCT04118374
Title: A Study to Determine Iatrogenic Hyperinsulinemia's Contribution to Insulin Resistance and Endothelial Dysfunction in Type 1 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Justin Gregory, Assistant Professor, Vanderbilt University Medical Center
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 190630
Record Dates: First submitted 2019-10-02; First posted 2019-10-08 (Actual); Results first posted 2025-10-28 (Actual); Last update posted 2025-10-28 (Actual); Status verified 2025-09

CONDITIONS: Diabetes Mellitus, Type 1
Keywords: low carbohydrate diet; hyperinsulinemia; insulin resistance; endothelial dysfunction; vascular health
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Hyperinsulinism; Insulin Resistance

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Carb Diet then Low Carb Diet (Experimental)
  Interventions: Other: Standard Carb Diet; Other: Low Carb Diet
- Low Carb Diet then Standard Carb Diet (Experimental)
  Interventions: Other: Standard Carb Diet; Other: Low Carb Diet

INTERVENTIONS:
Other: Standard Carb Diet — Approximately 50% of caloric intake will come from carbohydrate consumption.
Other: Low Carb Diet — Approximately 25% of caloric intake will come from carbohydrate consumption.

SUMMARY:
The investigators will test the hypothesis that reducing insulin doses using a low carbohydrate diet (LCD) will be associated with with improved insulin sensitivity (Aim 1) and blood vessel health (Aim 2).

DETAILED DESCRIPTION:
Insulin resistance (IR) is consistently found in patients with type 1 diabetes (T1DM) and pathophysiologically links T1DM with atherosclerotic disease. IR and nascent atherosclerosis, as characterized by endothelial dysfunction, are present early in T1DM. Although atherosclerosis leads to cardiovascular disease (CVD)-the predominant cause of death in T1DM-the early cardiometabolic processes driving atherosclerosis are not currently well-characterized. My overarching hypothesis is that IR and endothelial dysfunction in T1DM are, in part, iatrogenic, occurring as a function of nonphysiologic insulin delivery.

Previous research shows IR in T1DM is closely related to iatrogenic hyperinsulinemia. Iatrogenic hyperinsulinemia in T1DM results from injecting insulin into subcutaneous tissue rather than delivering insulin more physiologically into the hepatic portal vein. Hyperinsulinemia, per se, is closely linked with IR and independently predicts CVD in diabetic and nondiabetic populations. Thus, peripheral insulin delivery brings about unintended adverse cardiometabolic consequences in T1DM. The investigators propose a practical intervention to diminish iatrogenic hyperinsulinemia and thereby mitigate CVD risk. The investigators hypothesize that a reduction in iatrogenic hyperinsulinemia brought about by a low carbohydrate diet (LCD) will independently correlate with improved insulin sensitivity (Aim 1) and endothelial function (Aim 2).

In this pilot study, the investigators will mechanistically dissect the contribution of iatrogenic hyperinsulinemia to IR and endothelial dysfunction in 8 adults with T1DM using a crossover study of LCD vs. standard carbohydrate diet (SCD) to experimentally modify hyperinsulinemia. The investigators will quantify insulin sensitivity using hyperinsulinemic, euglycemic clamps and measure endothelium-dependent flow mediated vasodilation using high-resolution ultrasound.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18-60
* HbA1c: 5.6-9.0%
* Insulin delivery: must be on an insulin pump
* Glucose Monitor: must use a continuous glucose monitor (CGM)
* BMI 18-33 kg/m^2
* Body Mass >/= 50 kg ( 110 lbs)

Exclusion Criteria:

* severe hypoglycemia : >/= 1 episode in the past 3 months
* diabetes comorbidities (>= 1 trip to emergency department for poor glucose control in the past 6 months,
* New York Heart Association Class II-IV cardiac functional status
* SBP > 140 and DBP > 100 mmHg,
* eGFR by MDRD equation of <60 mL/min/1.73m^2
* AST or ALT > 2.5 times the upper limit of normal
* HCT <35%

medications

* any antioxidant vitamin supplement (<2 weeks before STUDY visit)
* any systemic glucocorticoid
* any antipsychotic
* atenolol, metoprolol, propranolol
* niacin
* any thiazide diuretic
* any OCP with > 35 mcg ethinyl estradiol,
* growth hormone
* any immunosuppressant
* any antihypertensive
* any antihyperlipidemic

other:

* pregnancy
* Tanner stage < 5
* peri or postmenopausal woman
* active smoker
* gluten-free diet requirement

Additional exclusion criteria for T1DM subjects

* any diabetes medication except insulin

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2021-11-24 (Actual); Primary Completion 2024-06-21 (Actual); Study Completion 2024-06-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Justin M Gregory, MD, MSCI, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: Yes
The datasets generated during and/or analyzed during the current study can be available from the corresponding author upon reasonable request. Data sets can be made available beginning 3 months and ending 5 years following article publication. No applicable resources have yet been generated or analyzed during the current study.
Supporting Information: Study Protocol, SAP, ICF, CSR

REFERENCES:
- [Result] Gregory JM, Smith TJ, Duffus SH, Brooks D, Akbar MN, Huntley MA, Gottlieb JA, LeStourgeon LM, Wilson CS, Beckman JA, Cherrington AD. A one-week reduced-carbohydrate diet to mitigate iatrogenic peripheral hyperinsulinemia does not improve insulin sensitivity or endothelial function in a randomized, crossover trial in patients with type 1 diabetes. Cardiovasc Diabetol. 2025 Mar 5;24(1):107. doi: 10.1186/s12933-025-02658-z. PMID 40045281

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 14 patients were screened for eligibility between November 2021 and March 2024. We recruited adults with type 1 diabetes (age 18-60 years, BMI 18-33 kg/m2, HbA1c 5.9-9.0%) from the Vanderbilt Eskind Diabetes Clinic and community sources in Nashville, TN.
Pre-assignment Details: In the full study, 14 participants enrolled and completed the screening visit. Two did not proceed past the run-in period due to scheduling conflicts and inconsistent nutrition logging.
Period: First Intervention (7 days)
Arm/Group | Standard Carb Diet then Low Carb Diet | Low Carb Diet then Standard Carb Diet
Started | 6 | 6
Completed | 6 | 6
Not Completed | 0 | 0
Period: Washout Period (21 days)
Arm/Group | Standard Carb Diet then Low Carb Diet | Low Carb Diet then Standard Carb Diet
Started | 6 | 6
Completed | 6 | 6
Not Completed | 0 | 0
Period: Second Intervention (7 days)
Arm/Group | Standard Carb Diet then Low Carb Diet | Low Carb Diet then Standard Carb Diet
Started | 6 | 6
Completed | 6 | 6
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Study Participants: Standard Carb Diet: Approximately 50% of caloric intake will come from carbohydrate consumption.
  Low Carb Diet: Approximately 25% of caloric intake will come from carbohydrate consumption.
  then all study participants crossed over to
  Low Carb Diet: Approximately 25% of caloric intake will come from carbohydrate consumption.
  Standard Carb Diet: Approximately 50% of caloric intake will come from carbohydrate consumption.
Arm/Group | All Study Participants
Number analyzed (Participants) | 12
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 33.9 [25.0 to 39.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 11
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 12
BMI [Median (Inter-Quartile Range); unit: kg/m^2] | 26.5 [21.7 to 28.4]
Weight [Median (Inter-Quartile Range); unit: kg] | 75.3 [66.8 to 92.0]
Height [Median (Inter-Quartile Range); unit: m] | 1.75 [1.68 to 1.88]
Waist-to-hip ratio [Median (Inter-Quartile Range); unit: ratio] | 0.83 [0.75 to 0.88]
HbA1c [Median (Inter-Quartile Range); unit: percentage of HbA1c] | 7.1 [6.7 to 7.7]
HbA1c [Median (Inter-Quartile Range); unit: mmol/mol] | 54 [49 to 61]
Type 1 diabetes duration [Median (Inter-Quartile Range); unit: years] | 20.5 [15.3 to 25.0]
Systolic blood pressure [Median (Inter-Quartile Range); unit: mmHg] | 120 [118 to 136]
Diastolic blood pressure [Median (Inter-Quartile Range); unit: mmHg] | 82 [78 to 90]
Heart rate [Median (Inter-Quartile Range); unit: bpm] | 65 [60 to 68]
Insulin analog used [Count of Participants; unit: Participants]
  Lispro | 6
  Aspart | 5
  Fast-acting insulin aspart | 1

OUTCOME MEASURES:

1. Primary Outcome: Change in Insulin Sensitivity Assessed as Glucose Infusion Rates
Description: Participants completed both a one-week RCD and a one-week SCD, separated by a three-week washout. After each intervention, we measured insulin sensitivity using a hyperinsulinemic-euglycemic clamp.To express GIR in mg of glucose per kg of fat-free mass per minute (mg/kg FFM/min), we divided the dextrose infusion rate by the fat-free mass determined by DEXA. Insulin sensitivity showed no significant difference between diets. GIR was 8.1 mg/kg FFM/min after the RCD and 8.6 mg/kg FFM/min after the SCD.
Time Frame: week 1 and week 5
Population: 12 participants received both interventions in this crossover study and were included in the analysis.
Measure: Median (Inter-Quartile Range); unit: mg/kg FFM/min
Arm/Group | Standard Carb Diet | Low Carb Diet
Number analyzed (Participants) | 12 | 12
mg/kg FFM/min | 8.6 [7.0 to 11.0] | 8.1 [6.7 to 10.1]
Statistical Analysis 1: Comparison: Standard Carb Diet vs Low Carb Diet; Test type: Superiority; p < 0.01, ANOVA; Median Difference (Final Values) = 0.2, 95% CI 2-sided [-0.5 to 1.8]

ADVERSE EVENTS:
Time Frame: through study completion, an average of 1 year
Description: Participants self-report
Arm/Group | Standard Carb Diet | Low Carb Diet
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 2/12 | 1/12
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard Carb Diet (N=12) | Low Carb Diet (N=12)
Headache (Nervous system disorders) | 2 (3) | 0 (0)
Shakiness (Nervous system disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-07-29): https://cdn.clinicaltrials.gov/large-docs/74/NCT04118374/Prot_SAP_001.pdf
  • Informed Consent Form (2022-07-14): https://cdn.clinicaltrials.gov/large-docs/74/NCT04118374/ICF_000.pdf